CLINICAL TRIAL: NCT04680299
Title: European Geriatric Emergency Departments Registry Study
Acronym: EGERS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gazi University (Other)
Collaborators: European Society for Emergency Medicine (EUSEM) Research Network (Network)
Responsible Party: Principal Investigator, Mehmet Akif Karamercan, Chair of Education and Fellowship Programme, Assoc. Prof., Gazi University
Other Study IDs: EUSEM-1
Record Dates: First submitted 2020-12-07; First posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Geriatric Patients; Emergencies; Length of Stay; Early Warning Score; Hospital Mortality
Keywords: Older Patients; Emergency Department; Early Warning Score
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Geriatric presentations to emergency services comprise a significant percentage of all emergency service presentations in Europe and it has been reported that 3-23% of all emergency service presentations from various regions of the countries. There are specific management practices for patients who are 65 years and older at emergency services. On the other hand several risk-scoring systems have been developed to define the severity class of the patient during their initial evaluation at emergency services.Only a few studies in the literature have evaluated risk-scoring systems for the geriatric patient group.Several studies have reported that risk-scoring systems, such as Identification of Seniors at Risk and Triage Risk Screening Tool, which are specifically developed for geriatric patients over 65 years who present to emergency services, are not sufficiently effective for evaluating patients in more severe conditions. Previously the TEDGeS (Turkish Emergency Departments Geriatric Scoring Study) pilot study was carried out and published by some of the investigators of this project.This pilot study enrolled all geriatric patients (age ≥ 65 years) and carried out in 13 centers from different cities of Turkey. This pilot study showed that geriatric patients not only constitute significant proportion of emergency department presentations but also these patients need more hospitalization. The predictive powers of the Modified Early Warning Score, Rapid Emergency Medicine Score and The Vital PAC Early Warning Score for hospitalization and mortality in geriatric patients those presented to emergency department are significantly high and might be concerned in the emergency department triage of these patients. Within the light of these pilot study results, the investigators have decided to execute this prospective, multinational, multicentric study with the main objective to determine the epidemiological and age related characteristics of geriatric patients presenting to the emergency department across Europe and evaluate early warning scoring systems systems regarding hospitalization, ICU admission and in-hospital mortality for geriatric patients.

DETAILED DESCRIPTION:
Due to improved prevention, diagnosis and treatment modalities, life expectancy worldwide has risen. The number of adults over 65 years of age who are presenting to emergency services is increasing in parallel with the prolongation of the average life expectancy. While geriatric presentations to emergency services comprise 40-50% of all emergency service presentations in the U.S., it has been reported that 3-23% of all emergency service presentations from various regions of the country comprise patients of 65 years of age and older. There are specific management practices for patients who are 65 years and older at emergency services due to the presence of co-morbidities and the change of physiological responses to acute diseases in advanced age.

Several risk-scoring systems have been developed to define the severity class of the patient during their initial evaluation at emergency services and generally named as Early Warning Scores. Early Warning Scores (EWS) incorporate physiological measurements, which do predict outcome although the addition of other simple clinical parameters might further improve the sensitivity and specificity of these scores. On the other hand all these EWS are simple and easy to calculate, making their use appropriate in an emergency setting. Of these EWS, the Modified Early Warning Score (MEWS), and the Rapid Emergency Medicine Score (REMS) have been widely used for many years (8) and The Vital PAC Early Warning Score (VIEWS) score was recently developed for the same purpose.

Only a few studies in the literature have evaluated risk-scoring systems for the geriatric patient group. Several studies have reported that risk-scoring systems, such as Identification of Seniors at Risk (ISAR) and Triage Risk Screening Tool (TRST), which are specifically developed for geriatric patients over 65 years who present to emergency services, are not sufficiently effective for evaluating patients in more severe conditions. Other studies have reported that the ESI triage classification predicts the prognosis correctly in only half of the patients over 65 years of age. In another study that evaluated the MEWS for the geriatric patient group, which was calculated during the presentation in emergency services, has been stated to have a prognostic value in terms of a poor result.

Previously the TEDGeS (Turkish Emergency Departments Geriatric Scoring Study) pilot study was carried out and published. This study enrolled all geriatric patients (age ≥ 65 years) and carried out in 13 centers (University Hospitals, Government Education and Research Hospitals and Military Hospital Emergency Departments) from different cities of Turkey.

Key findings were:

* Overall 30 % of hospitalized patients from Emergency Department (ED) are elderly patients and 30 % of these hospitalized patients were ICU hospitalizations
* In hospital mortality rate is about 6 % which is very high for general hospitalized patients
* The most common presenting symptoms are related to gastrointestinal systems and about 80 % of the cases using at least one chronic medication (22.2 % of the cases using more than 4 chronic medications
* About 45 % of the cases final diagnosis are related to cardiovascular system and gastrointestinal system and nearly 85 % of the hospitalized cases are treated in non-surgical clinics (cardiology-pulmonology-internal medicine 65 %)
* MEWS, VIEWS and REMS scores are significantly high in hospitalized patients compared to discharged from ED and also these three scores are high in ICU hospitalized patients compared to both ward hospitalized and discharged patients.
* MEWS, VIEWS and REMS scores are significantly high in non-survivors compared to survivors.
* MEWS, VIEWS scores has higher sensitivity and specificity in terms of in-hospital mortality

These results suggest that geriatric patients not only constitute significant proportion of ED presentations but also they need more hospitalization. The predictive powers of the MEWS, VIEWS and REMS scores for hospitalization and mortality in geriatric patients those presented to ED are significantly high and might be concerned in the ED triage of these patients.

Within the light of these results this multinational, multicentric, prospective, non interventional, observational study on geriatric patients presented to ED. The main objective is 'To determine Epidemiologic and Age Related Characteristics of Geriatric Patients presenting to the ED across Europe' and secondary objectives are 'To evaluate Early Warning Scoring systems (REMS, MEWS and VIEWS Scores) and determine most suitable Geriatric Emergency Medicine Risk Score regarding hospitalization, ICU admission and in-hospital mortality for patients; To determine the most effective triage elements that can be used to predict hospitalization of geriatric patients presented to ED; To determine the in hospital mortality and short term mortality rates of the patients above 65 years of age presenting to the ED across Europe; Sub analysis of ED discharged patients versus admitted patients for characteristics, comparison to recommended care and re-ED visit; Comparison of European data characteristics, investigation, treatment and outcome to similar data in other part of the world.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive geriatric patient presenting to the ED with any symptom
* 65 years or older

Exclusion Criteria:

* No acceptance to participated to the study
* End of life patients

Ages: 65 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients ≥ 65 years of age those presented to Emergency Departments with any symptom during the recruitment period of the study
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-02-21 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Medical history and co-morbidities | Baseline
  Listing of medical history and co-morbidities data provided by triage nurse, physician and the family during emergency department admission

SECONDARY OUTCOMES:
Length of Emergency Department stay | Up to 96 hours after registration to the ED
  Continuous outcome measured via the Patient Electronic Medical records defined in hours, measured from patient ED triage registration till discharged or hospitalized from ED.
Length of Hospital stay | 30 days after recruitment
  Continuous outcome measured via the Patient Electronic Medical records defined in Days, measured from admission to hospital wards or ICU date till discharge or death.
In Hospital Mortality | 30 days after recruitment
  Hospital mortality of geriatric patients admitted to hospital wards or ICU from emergency department

CONTACTS AND LOCATIONS:
Overall Officials: Said Laribi, MD., Principal Investigator — CHU Tours; Effie Polyzogopoulou, MD., Principal Investigator — University General Hospital ATTIKON; Kelly Janssens, MD., Principal Investigator — Unity Health Toronto; Anna Slagman, MD., Principal Investigator — UKSH Campus Kiel; Mehmet A. Karamercan, MD., Study Chair — Gazi University Faculty of Medicine; Zerrin D. Dundar, MD, Study Chair — Necmettin Erbakan University Meram Medicine Faculty
Locations (7):
- Clinical Hospital Sveti Duh, Zagreb, Croatia
- CHU Tours, Tours, France
- Charité Universitätsmedizin, Berlin, Duitsland, Germany
- University General Hospital ATTIKONi, Chaïdári, Griekenland, Greece
- St Michael's Hospital, Dublin, Ireland
- Turkey (Türkiye) (2):
  - Gazi University, Ankara
  - Necmettin Erbakan University Meram Medical Faculty, Konya

REFERENCES:
- [Background] Dundar ZD, Ergin M, Karamercan MA, Ayranci K, Colak T, Tuncar A, Cander B, Gul M. Modified Early Warning Score and VitalPac Early Warning Score in geriatric patients admitted to emergency department. Eur J Emerg Med. 2016 Dec;23(6):406-412. doi: 10.1097/MEJ.0000000000000274. PMID 25919485
- [Background] Cei M, Bartolomei C, Mumoli N. In-hospital mortality and morbidity of elderly medical patients can be predicted at admission by the Modified Early Warning Score: a prospective study. Int J Clin Pract. 2009 Apr;63(4):591-5. doi: 10.1111/j.1742-1241.2008.01986.x. Epub 2009 Feb 11. PMID 19220521
- [Background] Dundar ZD, Ayranci MK. Presenting symptoms of older emergency department patients: a single-center experience of 10,692 patients in Turkey. Acta Clin Belg. 2020 Dec;75(6):405-410. doi: 10.1080/17843286.2019.1655215. Epub 2019 Aug 12. PMID 31402765
- [Background] Lamantia MA, Stewart PW, Platts-Mills TF, Biese KJ, Forbach C, Zamora E, McCall BK, Shofer FS, Cairns CB, Busby-Whitehead J, Kizer JS. Predictive value of initial triage vital signs for critically ill older adults. West J Emerg Med. 2013 Sep;14(5):453-60. doi: 10.5811/westjem.2013.5.13411. PMID 24106542
- [Background] Buurman BM, van den Berg W, Korevaar JC, Milisen K, de Haan RJ, de Rooij SE. Risk for poor outcomes in older patients discharged from an emergency department: feasibility of four screening instruments. Eur J Emerg Med. 2011 Aug;18(4):215-20. doi: 10.1097/MEJ.0b013e328344597e. PMID 21317787
- [Background] Pines JM, Mullins PM, Cooper JK, Feng LB, Roth KE. National trends in emergency department use, care patterns, and quality of care of older adults in the United States. J Am Geriatr Soc. 2013 Jan;61(1):12-7. doi: 10.1111/jgs.12072. PMID 23311549
- [Background] Platts-Mills TF, Travers D, Biese K, McCall B, Kizer S, LaMantia M, Busby-Whitehead J, Cairns CB. Accuracy of the Emergency Severity Index triage instrument for identifying elder emergency department patients receiving an immediate life-saving intervention. Acad Emerg Med. 2010 Mar;17(3):238-43. doi: 10.1111/j.1553-2712.2010.00670.x. PMID 20370755
- [Background] Subbe CP, Kruger M, Rutherford P, Gemmel L. Validation of a modified Early Warning Score in medical admissions. QJM. 2001 Oct;94(10):521-6. doi: 10.1093/qjmed/94.10.521. PMID 11588210
- [Background] Wheeler I, Price C, Sitch A, Banda P, Kellett J, Nyirenda M, Rylance J. Early warning scores generated in developed healthcare settings are not sufficient at predicting early mortality in Blantyre, Malawi: a prospective cohort study. PLoS One. 2013;8(3):e59830. doi: 10.1371/journal.pone.0059830. Epub 2013 Mar 29. PMID 23555796

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-09-20): https://cdn.clinicaltrials.gov/large-docs/99/NCT04680299/Prot_SAP_ICF_000.pdf